CLINICAL TRIAL: NCT04651738
Title: Cell-free DNA Methylation for the Diagnosis and Monitoring of Endometrial Cancer: The Training and Validation Sets in China
Brief Title: Cell-free DNA Methylation for Endometrial Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lei Li (Other)
Responsible Party: Sponsor-Investigator, Lei Li, Professor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EC-METHY
Record Dates: First submitted 2020-11-26; First posted 2020-12-03 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Endometrial Cancer; Liquid Biopsy; DNA Methylation; Cervical Cytology; Diagnostic Accuracy; Training Set; Validation Set
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Intervention Model Description: All eligible patients accept DNA methylation testing in serum, cervical cytology and endometrial tissues.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): All eligible participants consenting to participate the study.
  Interventions: Diagnostic Test: DNA methylation testing

INTERVENTIONS:
Diagnostic Test: DNA methylation testing — Methylation testing of host DNA, namely, BHLHE22, CELF4, HAND2, and ZNF177

SUMMARY:
Liquid biopsy is challenging for the diagnosis of endometrial cancer. In this study, investigators perform the methylation testing of host DNA, namely, BHLHE22, CELF4, HAND2, and ZNF177, in the peripheral serum to discover the diagnostic and supervision roles of DNA methylation in endometrial cancer. The study compromises two stages.

In the training set, DNA methylation testing is performed in the endometrial tissues from patients with endometrial cancer and paired benign uterine lesions. The cut-off values of methylation are produced in this stage. On the meantime, DNA methylation testing is also performed in serum and in cervical cytology to reveal its accordance and accuracy compared with the results of endometrial tissues.

In the validation set, serum DNA methylation testing is performed in unselected patients with definite endometrial histology to validate its accuracy.

In training and validation sets, serum DNA methylation is also performed after major surgeries for endometrial cancer as to illustrate the changes of methylation testing, therefore, reflection the supervision role of DNA methylation.

ELIGIBILITY:
Inclusion Criteria:

* With definite histological diagnosis of endometrial cancer and paired benign uterine tumor in training set, and with definite histological diagnosis of uterine tumor in validation set.
* With sufficient fresh peripheral serum, cervical cytology, and endometrial samples for DNA methylation testing before with or without after major surgeries.
* Aged 18 years or older.
* Signed an approved informed consents

Exclusion Criteria:

* Not meeting all of the inclusion criteria.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2020-12-18 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Cut-off values of targeted DNA methylation in endometrial cancer | Two years
  The cut-off values are achieved by paired endometrial cancer and benign uterine tumor patients

SECONDARY OUTCOMES:
Accuracy of serum DNA methylation in endometrial cancer | Two years
  The accuracy is supported by sensitivity, specificity, negative predictive value and positive predictive value

CONTACTS AND LOCATIONS:
Overall Officials: Lei Li, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Lei Li, Beijing, Beijing Municipality, China